CLINICAL TRIAL: NCT01473225
Title: Can Calorie Labels Increase Caloric Intake? A Test of Possible Perverse Effects of Calorie Labels
Brief Title: Can Calorie Labels Increase Caloric Intake
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was pulled after unsuccessful pilot study
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, Principal Investigator, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P30AG034546 (NIH)
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Food Consumption

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Calorie label (Experimental)
  Interventions: Other: Calorie information
- No calorie label (Active Comparator)
  Interventions: Other: No calorie information

INTERVENTIONS:
Other: Calorie information — Nutrition label featuring calorie information will be provided.
  Arms: Calorie label
Other: No calorie information — No nutrition label will be provided in this condition.
  Arms: No calorie label

SUMMARY:
This study is a test of possible mechanisms by which calorie labels might lead people to increase calorie intake. The investigators hypothesize that calorie labels might increase calorie intake because 1) people infer that higher calorie foods are tastier, 2) calorie labels invoke thoughts of dieting, leading people to overconsume as a reaction, 3) people try to maximize calories consumed per dollar spent, and 4) calorie labels change one's goal motivation toward food, causing people to eat more.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to taste items used in study

Exclusion Criteria:

* Food allergies to items used in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09

PRIMARY OUTCOMES:
Calories consumed | At time of intervention (30 minutes)
  The investigators will assess how many calories are consumed by participants by weighing the cereal provided before and after participants complete the taste test portion of the study. This will happen within 30 minutes of the intervention, which is an experimental manipulation of whether or not calorie labels are present.

SECONDARY OUTCOMES:
Attitudes toward food | At time of intervention (30 minutes)
  Using survey measures, the investigators will assess how people feel toward the food item they just tasted, rating it in terms of perceived tastiness, healthiness, overall quality, and value. These ratings will be on a Likert scale from 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M VanEpps, BA, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States